CLINICAL TRIAL: NCT01860053
Title: A Behavioral Intervention to Decrease Vomiting and Improve Weight Loss in Post-Operative Laparoscopic Adjustable Gastric Banding (LAGB) Patients
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Tricia M. Leahey, Ph.D., Assistant Professor (Research), The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2030-09
Record Dates: First submitted 2013-05-06; First posted 2013-05-22 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Bariatric Surgery Complications
MeSH Terms: interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- behavioral intervention (Experimental)
  Interventions: Behavioral: behavioral intervention
- no treatment control (No Intervention)

INTERVENTIONS:
Behavioral: behavioral intervention — This intervention targets eating behavior to reduce vomiting and associated complications in post-operative LAGB patients.
  Arms: behavioral intervention

SUMMARY:
The purpose of this study is to reduce problematic vomiting and associated gastrointestinal symptoms in post-operative LAGB patients. We hypothesize that our behavioral intervention will yield greater reductions in vomiting and associated symptoms compared to our control condition.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70 years.
2. Received LAGB surgery with either a standard Lap-Band or a standard Realize Band.
3. Report vomiting at least 3x/week.
4. Agree to allow researchers to communicate with their surgeon regarding their care.
5. Fulfilled all hospital surgery criteria.

Exclusion Criteria:

1. Report a condition that in the judgment of the Principal Investigator would render them potentially unlikely to follow the protocol (e.g., major illness, plans to move out of the area, substance abuse or other significant psychiatric problems, organic brain disease).
2. Report planning to become pregnant during the time frame of the investigation.
3. Report a history of upper gastrointestinal dismotility.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-05; Primary Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
change in frequency of self-reported vomiting (number of vomiting episodes each week) measured via structured interview | baseline to week 6

SECONDARY OUTCOMES:
change in gastrointestinal symptom severity - questionnaire measures severity of various GI symptoms over the previous week and items are summed yielding an overall GI severity index | baseline to week 6

CONTACTS AND LOCATIONS:
Locations (1):
- Weight Control and Diabetes Research Center, Providence, Rhode Island, United States